CLINICAL TRIAL: NCT00913848
Title: A Single-Dose Comparative Bioavailability Study of Two Formulations of Divalproex Sodium 500 mg Delayed Release Tablets Under Fed Conditions
Brief Title: To Demonstrate the Relative Bioavailability of Divalproex Sodium 500 mg Delayed Release Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2005-1050
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-06

CONDITIONS: Epilepsy; Bipolar Disorder
Keywords: Treatment of Epilepsy and Bipolar Disorder
MeSH Terms: conditions — Epilepsy; Bipolar Disorder | interventions — Valproic Acid

ARMS (2):
- 1 (Experimental): Divalproex Sodium 500 mg DR Tablets (Sandoz Inc., USA)
  Interventions: Drug: Divalproex Sodium 500 mg DR Tablets (Sandoz Inc., USA)
- 2 (Active Comparator): Depakote 500 mg DR Tablets (Abbott Laboratories, USA)
  Interventions: Drug: Depakote 500 mg DR Tablets (Abbott Laboratories, USA)

INTERVENTIONS:
Drug: Divalproex Sodium 500 mg DR Tablets (Sandoz Inc., USA)
  Arms: 1
Drug: Depakote 500 mg DR Tablets (Abbott Laboratories, USA)
  Arms: 2

SUMMARY:
To demonstrate the relative bioavailability of Divalproex Sodium 500 mg delayed release tablets under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 21 Years to 47 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2005-10; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Xueyu (Eric) Chen, M.D., Principal Investigator — Pharma Medica Research, Inc.